CLINICAL TRIAL: NCT07373834
Title: Effects of Tirzepatide on Skeletal Muscle in Obesity
Brief Title: Tirzepatide and Muscle Outcomes in Obesity
Acronym: TIRMO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TIRMO-0120-121/2025-2711-6
Record Dates: First submitted 2025-12-05; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-11

CONDITIONS: Obesity (Disorder)
Keywords: Obesity; Tirzepatide; Skeletal muscle; Muscle quality; Muscle mass; Muscle strength; Muscle function; Myosteatosis; Muscle transcriptomics
MeSH Terms: conditions — Obesity | interventions — Tirzepatide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tirzepatide (Experimental)
  Interventions: Drug: Tirzepatide
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tirzepatide — Tirzepatide is a dual glucagon-like peptide-1 (GLP-1) and glucose-dependent insulinotropic polypeptide (GIP) receptor agonist. It will be administered via subcutaneous injection once weekly in a dose-titration scheme: starting at 2.5 mg and increased every 4 weeks by 2.5 mg up to a maximum of 15 mg, based on tolerability.
  Arms: Tirzepatide
Drug: Placebo — Placebo (saline solution) will be administered via subcutaneous injection once weekly with dose escalation following the same schedule (2.5 mg equivalent increments every 4 weeks) to preserve blinding integrity.
  Arms: Placebo

SUMMARY:
This study is evaluating whether a dual glucagon-like peptide-1 (GLP-1) and glucose-dependent insulinotropic polypeptide (GIP) receptor agonist, tirzepatide, can affect the function, structure and metabolism of skeletal muscles in adults with obesity. Participants, premenopausal females with obesity, will receive either tirzepatide or placebo over 24 weeks. Researchers will assess body weight, body composition, muscle strength and functional performance, neuromuscular function and will perform muscle biopsies before and after treatment to study molecular and histological changes following treatment. The goal of this study is to investigate the effects of tirzepatide on skeletal muscle function, quantity, quality and metabolism in adults with obesity as well as clarify the molecular and structural adaptations in skeletal muscle during tirzepatide-induced weight loss, addressing an important gap in understanding the impact of incretin-based therapies on muscle health.

ELIGIBILITY:
Inclusion Criteria:

* Female sex
* Age between 18 and 50 years
* BMI between 30 kg/m² and 40 kg/m²
* Stable body weight within the three months preceding study enrolment (defined as ≤ 5% change)
* No prior pharmacological or surgical interventions for obesity treatment
* Commitment to use barrier contraception and absence of plans for pregnancy within 8 months following enrolment

Exclusion Criteria:

* Sarcopenic obesity
* Pregnancy or lactation
* Postmenopausal status
* Diabetes
* Immobility
* Personal history of malignancy
* Personal history of pancreatitis
* Personal history of major depressive episodes
* Personal history of myopathy
* Personal or family history of medullary thyroid carcinoma
* Current treatment with metformin or systemic corticosteroids

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Change in Body Mass and Composition | Baseline to Week 24
  Measured primarily as changes in body weight and body composition measured by dual-energy X-ray absorptiometry (DXA).
Change in Quadriceps Muscle Strength | Baseline to Week 24
  Change in maximal knee extensor torque normalized to body mass (Nm/kg) will be evaluated using an isokinetic dynamometer.

SECONDARY OUTCOMES:
Change in MRI-derived Skeletal Muscle Composition and Myosteatosis | Baseline to Week 24
  Muscle volume and muscle fat fraction will be quantified using magnetic resonance imaging (MRI).
Change in Molecular Markers in Vastus Lateralis Muscle: Gene-level Differential Expression | Baseline to Week 24
  Transcriptome-wide RNA-sequencing will be performed on vastus lateralis muscle biopsies from all participants (depending on sample quality and RNA integrity) before and after the intervention to identify differentially expressed genes associated with tirzepatide treatment. Differential gene expression will be reported as log2 fold change (log2FC) between post and pre-intervention, derived from normalized RNA-sequencing read counts. Statistical significance will be summarized using false discovery rate (FDR)-adjusted p-values.
Change in Molecular Markers in Vastus Lateralis Muscle: Pathway-level Enrichment Analysis | Baseline to Week 24
  Pathway-level changes will be reported using normalized enrichment scores (NES) derived from gene set enrichment analysis (GSEA), together with false discovery rate (FDR)-adjusted q-values for biological processes including mitochondrial function, lipid metabolism, insulin signaling, inflammation, muscle atrophy, and myogenesis.
Change in Intramyocellular Lipid Content (IMCL) in Vastus Lateralis Muscle | Baseline to Week 24
  Assessed by Oil Red O staining using a standard protocol. IMCL will be quantified as the proportion of Oil Red O-positive area per fibre and averaged across available fibres per section per time point. Microscopy imaging and analysis settings will be kept consistent across time points, and assessors will be blinded to group/time.
Change in the Muscle Fiber Diameter of Type I and Type II Fibers | Baseline to Week 24
  Muscle fiber diameter will be measured on the biopsy section using routine light microscopy. Fiber typing (type 1 vs type 2) will be performed by standard immunohistochemistry for myosin heavy chain isoforms. The metric is mean minimal Feret diameter in micrometers, averaged across available fibers of same type.

OTHER OUTCOMES:
Change in Handgrip Strenght | Baseline to Week 24
  Change in maximal handgrip strength, normalized to body mass, will be assessed using a handheld dynamometer.
Changes in Lower-Limb Functional Performance | Baseline to Week 24
  Change in lower-limb functional performance assessed using standardized sit-to-stand testing.
Change in 6-Minute Walk Test (6MWT) | Baseline to Week 24
  The six-minute walk test (6MWT) will be used to assess functional exercise capacity. The outcome will be the total distance walked (meters) over 6 minutes on a flat corridor, following standardized guidelines.
Spatial Transcriptomics Analysis of Vastus Lateralis Muscle Biopsy Samples | Baseline to Week 24
  Potential exploratory: Feasibility-dependent analysis of spatial transcriptomic profiles in skeletal muscle biopsy. The objective is to identify treatment-related changes in spatial gene expression patterns in skeletal muscle tissue sections. A subset of approximately 8 patients (paired pre- and post-treatment muscle biopsy samples) will be selected for downstream analyses based on transcriptomic profiles obtained from the full RNA-seq dataset.
Electrophysiological Assessment of Motor Responses in Skeletal Muscles | Baseline to Week 24
  Potential exploratory: Electrophysiological recordings of motor responses (compound muscle action potentials, CMAP) will be assessed to evaluate potential changes in peripheral motor nerve excitability and neuromuscular function.

CONTACTS AND LOCATIONS:
Overall Officials: Mojca Jensterle Sever, Prof.MD, PhD, Principal Investigator — Department of Endocrinology, Diabetes and Metabolic Diseases, University Medical Centre Ljubljana
Locations (1):
- Department of Endocrinology, Diabetes and Metabolic Diseases, University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) to be shared will include demographic data, basic clinical measurements, body composition assessment, laboratory results, muscle strength and function assessment data, molecular data and histological features from skeletal muscle biopsies. All shared data will be fully de-identified, and no directly identifiable personal information will be included.